CLINICAL TRIAL: NCT02871375
Title: DAILIES TOTAL1® Multifocal Clinical Assessment in Challenging Patients
Brief Title: Clinical Assessment of DAILIES TOTAL1® (DT1) Multifocal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon, a Novartis Company (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CLE914-P001
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Results first posted 2017-11-24 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2017-10

CONDITIONS: Refractive Error
Keywords: myopia; presbyopia
MeSH Terms: conditions — Refractive Errors; Myopia; Presbyopia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DT1 MF, then Habitual (Other): Delefilcon A multifocal contact lenses in Period 1, followed by subject's habitual multifocal contact lenses in Period 2. Each product worn bilaterally (in both eyes) for 14 ± 3 days.
  Interventions: Device: Delefilcon A multifocal contact lenses; Device: Habitual multifocal contact lenses
- Habitual, then DT1 MF (Other): Subject's habitual multifocal contact lenses in Period 1, followed by delefilcon A multifocal contact lenses in Period 2. Each product worn bilaterally (in both eyes) for 14 ± 3 days.
  Interventions: Device: Delefilcon A multifocal contact lenses; Device: Habitual multifocal contact lenses

INTERVENTIONS:
Device: Delefilcon A multifocal contact lenses — Multifocal contact lenses worn in a daily wear, daily disposable modality (new pair of lenses each morning)
  Other Names: DAILIES TOTAL1® multifocal
Device: Habitual multifocal contact lenses — Multifocal contact lenses worn per subject's habitual prescription and habitual daily wear modality

SUMMARY:
The purpose of this study is to evaluate DAILIES TOTAL1® Multifocal (DTl MF) contact lenses in current multifocal contact lens wearers with symptoms of end of day discomfort compared to their habitual multifocal contact lens correction.

ELIGIBILITY:
Inclusion Criteria:

* Must sign an informed consent document;
* Current daily wearer of soft multifocal contact lenses for at least 6 months with symptoms of contact lens discomfort as defined by the prescreening Eligibility Questionnaire;
* Requires a near spectacle add of +0.50 to +2.50 diopters (D) (inclusive);
* Requires lenses within the power range of study lenses to be fitted;
* Best corrected VA (BCVA) of 20/30 (0.2 logarithmic minimum angle of resolution [logMAR]) or better in each eye at distance;
* Willing to wear study lenses for a minimum of 5 days per week, 6 hours per day, and attend all study visits;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any eye condition that contraindicates wearing contact lenses as determined by the Investigator;
* Any use of medications for which contact lens wear could be contraindicated, as determined by the Investigator;
* Monocular (only one eye functional) or fit with only 1 lens;
* Fitted with monovision;
* Prior refractive surgery (e.g., laser vision correction, photorefractive keratectomy, etc.);
* History of herpetic keratitis, ocular surgery, or irregular cornea;
* Currently wearing DT1 MF contact lenses;
* Other protocol-defined exclusion criteria may apply.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Manager, PLS, Study Director — Alcon, A Novartis Division

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 11 study centers located in the United States.
Pre-assignment Details: Of the 170 enrolled, 2 subjects were exited as screen failures prior to randomization. An additional 2 subjects were randomized in error but not exposed. This reporting group includes all randomized and exposed subjects (166).
Groups:
- DT1 MF / Habitual MF: Delefilcon A multifocal (MF) contact lenses in Period 1, followed by subject's habitual multifocal contact lenses in Period 2. Each product worn bilaterally (in both eyes) for 14 ± 3 days.
- Habitual MF / DT1 MF: Subject's habitual multifocal contact lenses in Period 1, followed by delefilcon A multifocal contact lenses in Period 2. Each product worn bilaterally (in both eyes) for 14 ± 3 days.
Period: Period 1, First 14 Days of Wear
Arm/Group | DT1 MF / Habitual MF | Habitual MF / DT1 MF
Started | 89 | 77
Completed | 89 | 76
Not Completed | 0 | 1
Not completed — Inclusion criteria not met | 0 | 1
Period: Period 2, Second 14 Days of Wear
Arm/Group | DT1 MF / Habitual MF | Habitual MF / DT1 MF
Started | 89 | 76
Completed | 89 | 76
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects who were exposed to any study lenses, except for lenses used for parameter optimization and fitting (Full Analysis Set).
Groups:
- Overall: Delefilcon A multifocal contact lenses and subject's habitual multifocal contact lenses worn bilaterally during Period 1 and Period 2 in a crossover assignment.
Arm/Group | Overall
Number analyzed (Participants) | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (5.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128
  Male | 38

OUTCOME MEASURES:

1. Primary Outcome: Binocular High Contrast/High Illumination (HC/HI) Visual Acuity (VA) at Intermediate Distance (80 cm)
Description: Visual Acuity (clarity or sharpness of vision) was measured at high contrast level. HC/HI VA was assessed binocularly (both eyes together) at 80 centimeters using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart and measured in logarithm of the minimum angle of resolution (logMAR). A lower logMAR value indicates better visual acuity.
Time Frame: Day 14, each product
Population: Full Analysis Set. Number Analyzed is the number of subjects with non-missing responses.
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- DT1 MF: Delefilcon A multifocal contact lenses worn bilaterally for 14 ± 3 days in Period 1 and Period 2
- Habitual MF: Subject's habitual multifocal contact lenses worn bilaterally for 14 ± 3 days in Period 1 and Period 2.
Arm/Group | DT1 MF | Habitual MF
Number analyzed (Participants) | 152 | 153
logMAR | -0.07 (0.10) | -0.09 (0.10)

2. Secondary Outcome: Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8) Score
Description: The abbreviated CLDEQ-8 is an 8-item questionnaire used to assess comfort and dryness. Total CLDEQ-8 score ranged from 0 to 37, where a lower score represented less symptomology.
Time Frame: Day 14, each product
Population: Full Analysis Set. Number Analyzed is the number of subjects with non-missing responses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | DT1 MF | Habitual MF
Number analyzed (Participants) | 165 | 165
units on a scale
  Period One: number analyzed (Participants) | 88 | 77
  Period One | 9.9 (5.4) | 17.0 (7.1)
  Period Two: number analyzed (Participants) | 77 | 88
  Period Two | 11.6 (6.3) | 13.0 (6.2)
  Overall | 10.7 (5.9) | 14.9 (6.9)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent for the duration of a subject's participation in the study (up to 44 days). AEs are reported as pre-treatment and treatment-emergent.
Description: An AE was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test article). AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator as outlined in the study protocol.
Groups:
- Pre-treatment: All subjects who consented to participate in the study prior to exposure to study lenses dispensed for 14-day wear
Arm/Group | Pre-treatment | DT1 MF | Habitual MF
All-Cause Mortality (participants affected / at risk) | 0/170 | 0/165 | 0/166
Serious Adverse Events (participants affected / at risk) | 0/170 | 0/165 | 0/166
Other Adverse Events (participants affected / at risk) | 0/170 | 0/165 | 0/166

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.